CLINICAL TRIAL: NCT03339011
Title: Effectiveness of Text Messages for Decreasing Inactive Behavior in Patients With Knee Osteoarthritis: a Pilot Randomised Controlled Study
Brief Title: Digital Motivation to Decrease Inactive Behaviour in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CB_IV
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS text message (Experimental): The content of the text messages is developed based on recommendation and advice from the Danish Health Authority about the importance of regular daily physical activity.
  For 6 weeks, the text messages will be send three times per week, twice during the week days and once in the weekend, based on previous experience with SMS as motivation for chronic pain patients.
  Interventions: Behavioral: Motivational SMS text message
- No intervention (No Intervention): No attention from the study

INTERVENTIONS:
Behavioral: Motivational SMS text message — Motivational text messages delivered to the participants' mobile phones. The text messages contain motivational text and advice on physical activity.
  Arms: SMS text message

SUMMARY:
Physical inactivity is a major risk behaviour with a potential for causing premature death, particularly among people with mobility limitations, such as knee osteoarthritis.

Digital motivational interventions (such as SMS) can motive to a healthy behaviour including increased physical activity.

The purpose of this study is to investigate if motivational text messages following an exercise intervention to improve mobility limitations will change the physical activity level in patients with knee osteoarthritis.

This study is designed as pilot randomized controlled trial, with equal randomization (1:1). Eligible participants will be randomised into one of two groups (intervention or control) after completing their baseline measurements. The intervention group will receive weekly motivational text messages and the control group will not receive any attention from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤18
* Diagnosed with knee osteoarthritis
* Owner of a smart phone or tablet
* Have just finished an exercise program for knee osteoarthritis

Exclusion Criteria:

* Not able to read and understand Danish
* Any condition, which in the opinion of the investigator would put the subject at increased safety risk by participation, or otherwise make the subject unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-07-29 (Actual); Study Completion 2018-07-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical inactivity | 6 weeks
  Physical inactivity is measured using an accelerometer based activity monitor. Physical activity is defined as time (in minutes) spent inactive, i.e. lying, sitting, standing during a day.

SECONDARY OUTCOMES:
Change form baseline in the Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks
  The Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire is used to assess patient reported outcomes on pain, function, and quality of life.
Transition questionnaire (TRANS-Q) of perceived change in knee symptoms | 6 weeks
  To investigate if participants experience a change in their osteoarthritis symptoms over time, they will be asked: "Pleas answer if you feel that your osteoarthritis symptoms have change for either the better, worse or no changes compared to before you entered this study" at the follow-up visit. The Participants can then check a box say: not change, a change for the worse or change for the better
Self-reported change in physical inactivity | 6 weeks
  At the follow-up visit participants will be asked "Have you changed your physical activity behaviour after completing the motivational intervention". This question will be asked at the end of the intervention period to investigate if the objective measurement of sedentary behaviour is related to the participants own perceived behaviour.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg University Hospitals, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bartholdy C, Bliddal H, Henriksen M. Effectiveness of text messages for decreasing inactive behaviour in patients with knee osteoarthritis: a pilot randomised controlled study. Pilot Feasibility Stud. 2019 Sep 7;5:112. doi: 10.1186/s40814-019-0494-6. eCollection 2019. PMID 31516729